CLINICAL TRIAL: NCT06277128
Title: A Phase 2 Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group, Dose-ranging Clinical Trial to Investigate the Efficacy and Safety of WS016 in the Patients With Hyperkalemia
Brief Title: A Study to Evaluate the Safety and Efficacy of WS016 in Patients With Hyperkalemia.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Waterstone Pharmaceutical (Wuhan) Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WS016-Ⅱ-01
Record Dates: First submitted 2024-02-03; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Hyperkalemia
MeSH Terms: conditions — Hyperkalemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- WS016 3g (Experimental)
  Interventions: Drug: WS016 3g
- WS016 6g (Experimental)
  Interventions: Drug: WS016 6g
- WS016 12g (Experimental)
  Interventions: Drug: WS016 12g
- Matching Placebo (Placebo Comparator)
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: WS016 3g — Acute treatment phase: WS016, oral, 3g , three times a day for 48 hours; Maintenance treatment phase: WS016, oral, 3g, once daily for 12 days.
  Arms: WS016 3g
Drug: WS016 6g — Acute treatment phase: WS016, oral, 6g , three times a day for 48 hours; Maintenance treatment phase: WS016, oral, 6g, once daily for 12 days.
  Arms: WS016 6g
Drug: WS016 12g — Acute treatment phase: WS016, oral, 12g , three times a day for 48 hours; Maintenance treatment phase: WS016, oral, 12g, once daily for 12 days.
  Arms: WS016 12g
Drug: Matching Placebo — Acute treatment phase: Matching Placebo, oral, three times a day for 48 hours; Maintenance treatment phase: Matching Placebo, oral, once daily for 12 days.
  Arms: Matching Placebo

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of different doses of WS016(3g, 6g and 12g) orally administered three times a day for 48 hours (acute treatment phase) vs placebo in the treatment of hyperkalemia, and to evaluate the efficacy of WS016(3g, 6g and 12g) orally administered once daily for 12 days ( maintenance treatment phase) vs placebo in maintaining normokalemia in participants have returned to normokalemia after the acute treatment phase.

DETAILED DESCRIPTION:
The study plan includes approximately 140 participants who will be randomly assigned to the WS016 and placebo treatment groups. Participants will begin a 48-hour acute treatment phase with three times-daily oral administrations. After the 48-hour acute treatment, participants have returned to normokalemia will be randomly assigned again to enter a 12-day maintenance treatment phase with once-daily oral administration.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years old, male or female;
2. The average blood potassium value measured by i-STAT for 2 consecutive times at screening is >5.0 mmol/L and ≤6.5 mmol/L (with an interval of 60±10 minutes between the 2 measurements);
3. Participants must provide informed consent for this trial, be able to maintain good communication with the investigator and comply with various requirements of the clinical trial (planned visits, laboratory tests, and other trial procedures, etc.).

Exclusion Criteria:

1. Pseudohyperkalemia, such as blood samples hemolysis caused by improper blood collection methods (e.g., tight tourniquet, excessive local massage, repeated clenching of the hand and release), participants with severe leukocytosis (>50×10^9/L) or thrombocytosis (>500×10^9/L);
2. Participants with hyperkalemia who require emergency treatment according to investigators assessment: e.g., with significant abnormalities on electrocardiogram (ECG) (e.g., flattened or absent P wave, widened QRS complex), or neuromuscular system symptoms;
3. Participants with symptomatic or uncontrolled atrial fibrillation, or asymptomatic persistent ventricular tachycardia (participants with controlled atrial fibrillation after drug treatment may be allowed to participate after assessment by the investigator);
4. Type 1 diabetes mellitus, or participants who developed diabetic ketoacidosis within 1 month before screening;
5. Participants with severe swallowing dysfunction, moderate to severe gastrointestinal dysfunction, or major gastrointestinal surgery (e.g., bariatric surgery or colectomy);
6. Participants who are receiving maintenance hemodialysis or peritoneal dialysis;
7. Participants who received sodium polystyrene sulfonate, calcium polystyrene sulfonate, patiromer sorbitex calcium, or sodium zirconium cyclosilicate within 3 days before the first administration of the study drug;
8. Participants who have undergone coronary artery bypass grafting, percutaneous interventional therapy (such as heart, cerebrovascular, aortic) or major surgeries including thoracic and cardiac surgery within 3 months prior to screening or are expected to undergo these procedures during the study period;
9. Participants who were hospitalized due to acute exacerbation of heart failure within 3 months before screening.
10. Participants who have undergone or are expected to undergo heart or kidney transplantation during the study period;
11. Participants with malignancies who are receiving antineoplastic treatment, or have uncontrolled systemic diseases or mental illnesses, and are evaluated by the investigators not suitable for participation in this study;
12. Participants with a life expectancy of less than 3 months;
13. Participants who test positive for HIV antibodies, syphilis antibodies, hepatitis C virus (HCV) antibodies, or hepatitis B surface antigen (HBsAg) with serum hepatitis B virus (HBV) -DNA ≥2000 IU/mL (only in HBeAg-positive patients) at screening;
14. Pregnant or breastfeeding women, or female participants who have had unprotected sexual intercourse within the past two weeks, or female participants who test positive for pregnancy; participants (or their partners) who have plans to conceive or donate sperm/ovum during the entire study period and 6 months after study completion, and are unwilling to use one or more contraceptive measures during the study period and 6 months after study completion.
15. Participants with any factors that are evaluated by the investigator, may affect the participant's ability to provide informed consent or comply with the study protocol, or may affect the trial results or participant safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2024-04-18 (Estimated); Study Completion 2024-08-04 (Estimated)

PRIMARY OUTCOMES:
Exponential rate of change in serum potassium(S-K) levels during the acute treatment phase | Through the initial 48-hour acute treatment phase (from baseline to hour 48)
Exponential rate of change in S-K levels during the maintenance treatment phase | Through 12 days of maintenance treatment phase (from Day 3 to Day 15)

SECONDARY OUTCOMES:
Mean change in S-K levels during the acute treatment phase | Through the initial 48-hour acute treatment phase
  The mean change in S-K levels during the acute treatment phase compared to baseline
Proportion of participants recover from hyperkalemia | Through the initial 48-hour acute treatment phase
  The percentage of participants whose S-K levels return to normal during the acute treatment phase
Time to normalization in S-K levels | Through the initial 48-hour acute treatment phase
  The time(hours) it takes for participants' S-K levels to return to normal during the acute treatment phase
Proportion of patients remaining normokalemic | Day 15
  The percentage of participants whose S-K levels remain within the normal range (3.5-5.0 mmol/L) at the end of the maintenance treatment phase
Mean change in S-K levels during the maintenance treatment phase | Through 12 days of maintenance treatment phase (from Day 3 to Day 15)
  The mean change in S-K levels during the maintenance treatment phase compared to baseline

CONTACTS AND LOCATIONS:
Locations (26):
- China (26):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Peking University Shougang Hospital, Beijing, Beijing Municipality
  - Zhongshan Hospital, Xiamen University, Xiamen, Fujian
  - The Affiliated Hospital of Hebei University, Baoding, Hebei
  - Hebei Traditional Chinese Medicine Hospital, Shijiazhuang, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Hospital of Qiqihar, Qiqihar, Heilongjiang
  - The First People's Hospital of Nanyang City, Nanyang, Henan
  - Puyang Oilfield General Hospital, Puyang, Henan
  - Shiyan Taihe Hospital, Shiyan, Hubei
  - Wuhan No.4 Hospital, Wuhan, Hubei
  - Zhuzhou Central Hospital, Zhuzhou, Hunan
  - Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Sir Run Run Hospital, Nanjing Medical University, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Shenyang Central Hospital, affiliated to Shenyang Medical College, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - The First People's Hospital of Tancheng County, Linyi, Shandong
  - Qilu Hospital of Shandong University (Qingdao), Qingdao, Shandong
  - Minhang District Central Hospital, Shanghai, Shanghai Municipality
  - Shanghai First People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai No.5 Hospital, Shanghai, Shanghai Municipality
  - Shanghai Tongji Hospital, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Undecided